CLINICAL TRIAL: NCT01771094
Title: Effect of Sweetness of the Beverage in Thirst Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Pedro Miguel Fernandes Ramos de Carvalho, Invited Assistant, Universidade do Porto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IHS/FCNAUP-002; Nº30/CEUP/2011
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Thirst

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (placebo) - Water (Placebo Comparator): This group will drink water in 1st trial
  Interventions: Behavioral: Effect of sweetness of the beverage in thirst sensation
- Group 3 (Intervention) - "Low" Sucralose (Experimental): This group will drink Decarbonized Pineapple with a 50% decrease of sucralose face to standard beverage in 1st trial
  Interventions: Behavioral: Effect of sweetness of the beverage in thirst sensation
- Group 2(Intervention)-"High" Sucralose (Experimental): This group will drink Decarbonized Pineapple Diet Soda with a 50% increase of sucralose face to standard beverage in 1st trial
  Interventions: Behavioral: Effect of sweetness of the beverage in thirst sensation

INTERVENTIONS:
Behavioral: Effect of sweetness of the beverage in thirst sensation — Effect of sweetness of the beverage in thirst sensation:
  The participants will drink Water (control group),"High Sucralose" - Decarbonized Pineapple Diet Soda with a 50% increase of sucralose face to standard beverage, and "Low Sucralose" - Decarbonized Pineapple with a 50% decrease of sucralose face to standard beverage. The beverages will be presented chilled but without ice in 500 ml portions in opaque plastic containers and participants will be asked to consume the entire amount within 15 min.

SUMMARY:
The purpose of this study is to determine if water and diet soft drinks with different levels of sweeteners have the same effect on thirst.

DETAILED DESCRIPTION:
Participants should be in the laboratory at 8.00 in order to collect the values of weight, height, total body water, intracellular water and extracellular water in a Segmental Multi Frequency Body Composition Monitor (TANITA MC 180 MA®). Then, a blood sample will be collected for analysis of blood glucose and osmolality. They will sit at individual tables for the duration of the session and were allowed to read, listen to music with earphones, or use their portable computers with the exception of internet access to minimize visual cues (e.g., unwanted publicity for beverages or visiting Web sites showing pictures of food and drinks), which may have effect on thirst. Breakfast will be served at 9.30 on every occasion and preload stimuli will be offered exactly 60 minutes after breakfast (at 10.30). Lunch will be provided at 13.00. Motivational ratings will be first obtained at the end of collection of blood sample (baseline or time 0) and every 30 minutes thereafter until the lunch time (times 1 through 7). After lunch (time 8), participants will complete the last set of ratings and will bring a food diary to record all food and fluid intake until 00.00 that day.

ELIGIBILITY:
Exclusion Criteria:

* pregnant and nursing women
* smokers
* athletes
* subjects under medication(except oral contraceptives in women)

Inclusion Criteria:

* body mass index(BMI) between (18,5 - 27,5 kg/m2)
* regular consumers of breakfast
* stable in weight for the past 6 months
* not dieting to gain or lose weight
* like all drinks and food available in study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Motivational Ratings | 1 day
  Participants will rate their hunger, thirst, nausea, mouth dryness, desire to eat, desire to drink using nine point category scales. The unipolar adjective scales were anchored at each end with labels: 1 = not at all and 9 = extremely. Participants also rated their perception about beverage sweetness along nine point hedonic preference scales where 1 = no sweet at all and 9 = extremely sweet

SECONDARY OUTCOMES:
Food Behavior After Intervention | 1 day
  After lunch, participants will bring a food diary to record all food and fluid intake until 00.00 that day. Then, we will analyse total calories ingested, total fluid ingested and the volume of sugar and sugary beverages ingested.
Physiological Parameters | 1 day
  Glycaemia, blood osmolality and hydration parameters (total body water, intra and extracellular body water) will be assessed before and after the ingestion of beverages
Amount of water ingested | 1 day
  After the ingestion of 3 preloads with the beverages in study, the participants will lunch the same meal with free water ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Pedro R Carvalho, PhD Student, Principal Investigator — FCNAUP
Locations (1):
- Faculty of Nutrition and Food Sciences - University of Porto, Porto, Porto District, Portugal